CLINICAL TRIAL: NCT01938872
Title: Evaluating the Effectiveness of Paclitaxel-eluting Balloons for Below-the-knee Angioplasty in Patients With Critical Limb Ischemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Leonardo Bolognese, MD, Director, Ospedale San Donato
Other Study IDs: Arezzo010
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Critical Limb Ischemia
Keywords: critical limb ischemia; drug-eluting balloon; restenosis
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PEB angioplasty: paclitaxel eluting balloon angioplasty in below-the-knee lesions
  Interventions: Procedure: paclitaxel eluting balloon angioplasty in below-the-knee lesions

INTERVENTIONS:
Procedure: paclitaxel eluting balloon angioplasty in below-the-knee lesions
  Other Names: FREEWAY™ (Eurocor GmbH)

SUMMARY:
to evaluate the the effectiveness of paclitaxel-eluting balloon for below-the-knee angioplasty in terms of restenosis at 12 months

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* angiographic stenosis>50% or occlusion of one below-knee vessel

Exclusion Criteria:

* allergy to Paclitaxel
* contraindication for combined antiplatelet treatment
* life expectancy <1 year
* hypersensitivity or contraindication to one of the study drugs
* lack of consent
* need for amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing below-the-knee angioplasty with paclitaxel eluting balloon for critical limb ischemia
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
angiographic binary restenosis | 12 months
  incidence of binary restenosis

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Department, Ospedale S.Donato, Arezzo, AR, Italy